CLINICAL TRIAL: NCT03314259
Title: Prophylactic Alpha-blockers in the Prevention of Post-operative Urinary Retention After Inguinal Hernia Repair: A Randomized Double-Blind Placebo-Controlled Trial
Brief Title: Prophylactic Alpha-blockers in the Prevention of Urinary Retention Post Inguinal Hernia Repair
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016/00295-SRF0001
Record Dates: First submitted 2017-09-05; First posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Urinary Retention; Inguinal Hernia
MeSH Terms: conditions — Urinary Retention; Hernia, Inguinal | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double blind, placebo- controlled trial. After establishing the eligibility of the patients and obtaining the necessary informed consent, the research assistant (third party) will provide them with pre-assigned sealed envelopes that contain information with regards to their designated arm. The patients in the intervention arm will then be provided with Tamsulosin, while the rest will be given the placebo in a similar packaging. Blinded personnel would include the study participants and doctors/nurses involved in the surgery and peri-operative care. As such, participants, care providers and outcome assessors would all be blinded in our study. There will be no unmasking in our trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamsulosin (Experimental): Patients will then consume oral tamsulosin 0.4mg every morning daily for 5 days prior to elective surgery
  Interventions: Drug: Tamsulosin
- Placebo (Placebo Comparator): Patients will then consume placebo every morning daily for 5 days prior to elective surgery
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Tamsulosin — Tamsulosin is a alpha blocker and has a good safety profile that has been used extensively in Urological patients. Potential safety issues would include a minimal risk of orthostatic hypotension and hypersensitivity reaction to tamsulosin in our study population
  Arms: Tamsulosin
Drug: Placebo Oral Tablet — placebo is a tablet made to mimic tamsulosin tablet with same size and colour with no active ingredient
  Arms: Placebo

SUMMARY:
Post operative urinary retention ( POUR) is caused by sympathetic activation of the internal urethral sphincter after surgery. The smooth muscles of the around the internal urethral sphincter have been demonstrated to be rich in alpha-1 adrenergic receptors. Our research idea is novel because there has been no prior prospective study conducted using alpha-blockers to reduce post-operative urinary retention in patients undergoing inguinal hernia repair. The proposed research is important as existing studies that sought to understand POUR have merely established the risks factors involved. Despite so, the incidence of POUR remains high and no studies to date have investigated the use of specific interventions to reduce the risk of POUR.

This is essential as patients who develop POUR have also been successfully shown to have significantly longer length of hospitalisation. Besides, the development of POUR can also cause significant pain/discomfort, increase risks of long-term urethral catheterisation and predispose patients to urinary tract infections

DETAILED DESCRIPTION:
The study will be conducted as a randomised, double blind, placebo-controlled trial. This is a single center trial. The experimental design and procedure will be performed in accordance to the CONSORT guidelines. Patients will be assessed for eligibility, and selected based on the inclusion and exclusion criteria. Once eligible, informed consent will be obtained for every patient, and those in agreement to the participation of the trial will be randomly provided with pre-assigned sealed envelopes containing either tamsulosin or placebo, for which patient and investigators will be blinded to. Patients will then consume either oral tamsulosin 0.4mg or placebo daily for 5 days prior to elective surgery. A baseline postural blood pressure measurement will be taken before and after the 1st dose, and patients will be informed to look out for symptoms of hypersensitivity reactions and orthostatic hypotension, and to cease consumption should they develop. Prior to surgery, the patients will require to report to the study team if they had finished all 5 drug doses. Patients who develop intercurrent illnesses or have urgent matters at hand that would require their surgery to be postponed will receive another 5 drug doses that is to be consumed prior the their next scheduled surgical date. During the surgery, a maximum dose of 0.1mg/kg of morphine can be given to patients. No ilioinguinal block will be performed for patients, but local anesthesia 10mls 0.5% Bupivacaine will be infiltrated into the wound sites. The patients will then be monitored in the 23 hour short stay ward, during which the patient's wound site, scrotum, pain levels and ability to pass urine will be assessed prior to being discharged. All patients will be provided with a maintenance drip post operatively. Patients will also be placed on paracetamol 1g 6 hourly strictly and tramadol 50mg 8 hourly as per required. Alternative analgesia will be provided should patients have existing allergies to these drug classes.

Patients will be assessed for presence of voiding difficulty 6 hours post operatively, and patients who complain of voiding difficulty or inability to pass urine within 6 hours post operatively will be defined to have POUR, while a bladder scan will be performed will be performed . Patients with existing bladder volume of more than 400mls will be catheterised, while those with less than 400mls will be followed up with subsequent 2 hourly bladder scans, and catheterised should their bladder volume be beyond 400mls. Once discharged, patients will receive a phone call at 24 hours post discharge and scheduled to return for a follow up appointment 1 weeks later in the clinic where urinary symptoms will once again be assessed in both settings. The end points of incidence of POUR/catheterisation, length and cost of hospitalisation, rates of same day discharge, and patient satisfaction in both arms will be recorded and analysed. Patients will be analysed via an intention to treat basis, and patients who defaulted treatment (did not receive full 5 doses of medicine), did not turn up for surgery or lost to subsequent follow up post operatively will be taken into account, and reported and analysed accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Males of 41 to 80 years old who are going for elective inguinal hernia repair (laparoscopic or open) under general anesthesia.

Exclusion Criteria:

Patient whom has any of the following will be excluded:

* Contraindication to tamsulosin : known allergy, known orthostatic hypotension, significant cardiac co-morbidities ( New york heart association functional classification >2) or heart failure
* End stage renal failure
* More than two anti-hypertensive use/long term alpha blockers/beta blockers/anticholinergic (eg : buscopan)
* Previous urological or pelvic surgery
* Known benign prostatic hyperplasia on medications
* Long term indwelling catheters
* Concurrent neurologic disease such as stroke, poliomyelitis, cerebral palsy, multiple sclerosis, spinal lesions, diabetic and alcoholic neuropathy

Ages: 41 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 300 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Post operative urinary retention | 6 hours post surgery
  patients who complain of voiding difficulty or inability to pass urine within 6 hours post operatively will be defined to have POUR, while a bladder scan will be performed . Patients with existing bladder volume of more than 400mls will be catheterised, while those with less than 400mls will be followed up with subsequent 2 hourly bladder scans, and catheterised should their bladder volume be beyond 400mls.

CONTACTS AND LOCATIONS:
Overall Officials: Lomanto Davide, MD, PhD, FAMS, Principal Investigator — National University of Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No